CLINICAL TRIAL: NCT00203489
Title: A Prospective Randomized Double-Blind Trial of a Polyhexamethylene Biguanide (PHMB) Impregnated Gauze Dressing for the Prevention of Chronic Wound Colonization With Resistant and Prevalent Microorganisms
Brief Title: A Clinical Study of An Antimicrobial Gauze Dressing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Reallocation of funding.
Sponsor: Tyco Healthcare Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Study Protocol 331.18
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-11

CONDITIONS: Wounds
MeSH Terms: conditions — Wounds and Injuries

INTERVENTIONS:
Device: KERLIX A.M.D. Gauze

SUMMARY:
The purpose of this study is to determine if a new antimicrobial gauze dressing is better than the current method of dressing open wounds with plain sterile gauze. It is hoped that the antimicrobial gauze will reduce the number of germs in the open wound and even improve the rate of healing.

DETAILED DESCRIPTION:
Without adequate debridement, chronically infected wounds persist and form a nidus for the acquisition of antimicrobial-resistant microorganisms. Multiple studies state that patients with chronic wounds were colonized with one or more resistant bacteria, and that the presence of a chronic wound or decubitus ulcer was associated with a statistically increased likelihood of colonization with methicillin-resistant Staphylococcus aureus (MRSA), ciprofloxacin-resistant gram-negative bacilli (GNB),colonization and infection with ceftazidime-resistant Escherichia coli and Klebsiella pneumoniae.

Recently, a newly formulated gauze dressing impregnated with an antiseptic agent has become available. This product offers the promise of a combined benefit of wet-to-dry mechanical debridement, while providing high local concentrations of a potent antiseptic to prevent colonization and infection of the wound by resistant microorganisms, potentially enhancing wound healing.

This study proposes to determine if use of the antimicrobial gauze in routine wound care results in a lower rate of chronic wound colonization with resistant microorganisms and prevalent microorganisms as compared to standard wound care (with non-antimicrobial gauze).

ELIGIBILITY:
Inclusion Criteria:

1. The subject is receiving care at the study wound care clinics.
2. The subject is 18 years of age or older.
3. The subject or authorized representative has signed the Informed Consent form.
4. The subject has a chronic wound as a result of pressure ulceration (grade III and IV ulcers only), underlying vascular disease ("leg ulcer"), diabetes mellitus (grade 2 and 3 ulcers only), or recent surgery.

Exclusion Criteria:

1. The subject has a chronic ulcer that is a result of a condition other than that defined in the inclusion criteria.
2. The subject has stage I and II pressure ulceration.
3. The subject has a superficial (grade 0 or 1) or limb-threatening diabetic foot ulceration (grade 4 or 5).
4. The subject has a leg ulcer related to carcinoma.
5. The subject is scheduled to go for amputation or surgical flap procedure as a result of an open wound.
6. Subject is scheduled to receive a V.A.C.® (Vacuum Assisted Closure) Dressing [V.A.C.® (Vacuum Assisted Closure) Dressing KCI, Kinetic Concepts, Inc., San Antonio, TX].
7. The subject has extensive burns or another acute diffuse skin condition (Stevens-Johnson Syndrome).
8. The subject has a history of hypersensitivity to Chlorhexidine Gluconate (CHG) or Polyhexamethylene Biguanide (PHMB).
9. The subject has severe systemic infection characterized by the systemic inflammatory response syndrome.
10. The subject has taken part in a wound healing study within the past month.
11. The subject has suspected or confirmed underlying osteomyelitis contiguous to the ulcer and is not receiving systemic antimicrobial therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-06; Study Completion 2007-08

PRIMARY OUTCOMES:
Rate of chronic wound colonization with resistant/prevalent microorganisms.

SECONDARY OUTCOMES:
Rate of wound surface area healing over time; Antibiotic utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya M. Eggleston, RN, MPH, Study Director — Tyco Healthcare/Kendall
Locations (1):
- Sunnybrook & Women's College Health Sciences Centre, Toronto, Ontario, Canada